CLINICAL TRIAL: NCT03133845
Title: Shaping Anesthetic Techniques to Reduce Post-Operative Delirium
Acronym: SHARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Mercy Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00113655
Record Dates: First submitted 2015-10-23; First posted 2017-04-28 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Delirium; Lumbar Radiculopathy; Lumbar Osteoarthritis; Lumbar Spine Disc Degeneration
Keywords: delirium; elderly; lumbar; surgery
MeSH Terms: conditions — Delirium; Radiculopathy; Osteoarthritis, Spine | interventions — Propofol; Neoadjuvant Therapy; Analgesia; Fentanyl; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- General anesthesia (Active Comparator): In this group patients will receive general anesthesia. Anesthetic induction will occur with propofol (generally 1-2 mg/kg), maintenance with a volatile anesthetic, muscle paralysis with a muscle relaxant, and pain control with fentanyl (generally 2-5 mcg/kg titrated). Patients on baseline opioids may receive additional opioids (such as dilaudid) based on clinical criteria. The anesthetic provider will be blinded to BIS values. Discretionary use of intrathecal morphine may be used.
  Interventions: Procedure: Induction with propofol; Procedure: Maintenance anesthetic using a volatile anesthetic; Procedure: Muscle relaxant during maintenance anesthesia; Procedure: Pain control with fentanyl; Procedure: Bispectral Index (BIS) monitoring for depth of anesthesia; Procedure: Cerebrospinal fluid collection; Procedure: Administration of intrathecal morphine
- Spinal anesthesia with light sedation (Experimental): In this group patients will receive light sedation with propofol and a spinal anesthetic. Spinal anesthesia will be obtained by injecting approximately 10-15 mg of bupivacaine into the subarachnoid space. Up to 2 mg of midazolam may be given during spinal needle insertion. Although spinal anesthesia is sufficient for surgery, sedation is routinely administered using a propofol infusion, titrated to a BIS>60-70. Discretionary use of intrathecal morphine may be used.
  Interventions: Procedure: Light sedation with propofol; Procedure: Bispectral Index (BIS) monitoring for depth of anesthesia; Procedure: Spinal Anesthesia; Procedure: Midazolam administered during spinal anesthesia; Procedure: Cerebrospinal fluid collection; Procedure: Administration of intrathecal morphine

INTERVENTIONS:
Procedure: Light sedation with propofol — Patients having lumbar spinal surgery and receiving spinal anesthesia will receive propofol for light sedation.
  Arms: Spinal anesthesia with light sedation
Procedure: Induction with propofol — Patients having lumbar spinal surgery and receiving general anesthesia will receive propofol and their induction agent.
  Arms: General anesthesia
Procedure: Maintenance anesthetic using a volatile anesthetic — Patients having lumbar spinal surgery and receiving general anesthesia will receive a volatile anesthetic for their maintenance anesthesia.
  Arms: General anesthesia
Procedure: Muscle relaxant during maintenance anesthesia — Patients having lumbar spinal surgery and receiving general anesthesia with receive a muscle relaxant for muscle paralysis.
  Arms: General anesthesia
Procedure: Pain control with fentanyl — Patients having lumbar spinal surgery and receiving general anesthesia will receive fentanyl for their pain during surgery.
  Arms: General anesthesia
Procedure: Bispectral Index (BIS) monitoring for depth of anesthesia — All patients will be monitored with Bispectral Index (BIS) to monitor the patient's depth of anesthesia.
Procedure: Spinal Anesthesia — Patients receiving spinal anesthesia will receive bupivacaine into the subarachnoid space.
  Arms: Spinal anesthesia with light sedation
Procedure: Midazolam administered during spinal anesthesia — Midazolam may be administered during spinal needle insertion for patients receiving spinal anesthesia.
  Arms: Spinal anesthesia with light sedation
Procedure: Cerebrospinal fluid collection — 8 ml of cerebrospinal fluid may be collected prior to the administration of intrathecal administration of morphine for pain control.
Procedure: Administration of intrathecal morphine — Patient may receive intrathecal morphine for post-operative pain control.

SUMMARY:
The purpose of this study is to determine if light sedation with spinal anesthesia reduces the incidence of delirium compared to receiving general anesthesia during spinal surgery in older adults.

DETAILED DESCRIPTION:
Post-operative delirium is a common occurrence in older adults. Post -operative delirium has been associated with cognitive decline after hospitalization. Developing perioperative management strategies to prevent delirium may also reduce potential cognitive decline in older adults after surgery. The choice and dose of anesthetic and sedative drugs are known risk factors in the development of delirium. Excessive doses of anesthetic and sedation drugs during surgery have been associated with poor outcomes that occur after surgery. Currently depth of anesthesia can be measured by an additional monitoring technique called Bispectral Index (BIS).

The purpose of this study is to determine if light sedation with spinal anesthesia reduces the incidence of delirium compared to receiving general anesthesia during spinal surgery in older adults. Previous studies have shown that using light sedation and spinal anesthesia during surgery may reduce the incidence of delirium up to 50%.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age 65 and over.
* Patients undergoing lumbar fusion performed by Dr. Charles Edwards II, Dr. Charles Edwards, Dr. Clayton Dean , or Dr. Justin Park at Mercy Medical Center.
* Expected length of surgery <3 hours.
* Ability to understand study procedures and to comply with them for the entire length of the study

Exclusion Criteria:

* Contradictions to spinal anesthesia (severe aortic stenosis, anti-coagulant or antiplatelet medications, other)
* Body mass index > 40 kg/m2
* prior lumbar fusion from L2-L5 in entirety
* Communication issues precluding delirium assessment or sedation
* Dementia or mini-mental status exam score < 24
* Psychiatric disease that would preclude cooperation with sedation with spinal anesthesia
* Any other reason that the attending anesthesiologist or surgeon feels that clinical circumstances dictate a strong preference for either spinal or general anesthesia.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium | First 3 postoperative days
  The patient will be assessed for delirium using the Confusion Assessment Method on each of the first 3 post-operative days.

SECONDARY OUTCOMES:
Assessment of cognitive status at 3 months using the Verbal Fluency Test | 3 months after surgery
  The participant will be administered the Verbal Fluency Test to measure verbal fluency. Participants are given 1 minute to name as many words as possible beginning with a letter. Participants are then given 1 minute to name as many words as possible beginning with a different letter. Participants are then given 1 minute to name as many words as possible in a category. The score is the total number of different words produced for all 3 trials and will be compared to the score obtained at baseline.
Assessment of cognitive status at 1 year using the Verbal Fluency test. | 1 year after surgery
  The participant will be administered the Verbal Fluency Test to measure verbal fluency. Participants are given 1 minute to name as many words as possible beginning with a letter. Participants are then given 1 minute to name as many words as possible beginning with a different letter. Participants are then given 1 minute to name as many words as possible in a category. The score is the total number of different words produced for all 3 trials and will be compared to the score obtained at baseline.
Assessment of functional status at 3 months using the Instrumental Activities of Daily Living (IADL) test. | 3 months after surgery
  At 3 months, the participant's functional status will be assessed using the instrumental activities of daily living (IADL) scales. Scores can range from 0-14 with 14 being high functioning and 0 being low functioning. This score will be compared to the baseline score.
Assessment of functional status at 1 year using the Instrumental Activities of Daily Living (IADL) test. | 1 year after surgery
  At 1 year, the participant's functional status will be assessed using the instrumental activities of daily living (IADL) scales. Scores can range from 0-14 with 14 being high functioning and 0 being low functioning. This score will be compared to the baseline score.
Assessment of functional status at 3 months using the Short Form 12 Health Survey (SF-12) | 3 months after surgery
  This is a survey that measures the patient's own self reported view on their health. Scores range from 0-100, with 0 indicating the lowest level of health and 100 indicating the highest level of health.
Assessment of functional status using at 1 year the Short Form 12 Health Survey (SF-12) | 1 year after surgery
  This is a survey that measures the patient's own self reported view on their health. Scores range from 0-100, with 0 indicating the lowest level of health and 100 indicating the highest level of health.
Assessment of functional status at 3 months using the Oswestry Disability Index (ODI) | 3 months after surgery
  This survey measures self-reported disability due to low pain. Scores range from 0-100, with 0 being minimal or no disability and 100 being severe disability. This score will be compared to the baseline score.
Assessment of functional status at 1 year using the Oswestry Disability Index (ODI) | 1 year after surgery
  This survey measures self-reported disability due to low pain. Scores range from 0-100, with 0 being minimal or no disability and 100 being severe disability. This score will be compared to the scores obtained at baseline and 3 months after surgery.
Assessment of cognitive status at 3 months using Trail Making Test | 3 months after surgery
  This test provides information visual search speed, scanning, speed of processing, mental flexibility, and executive functioning. The test is scored by the amount of time it takes to complete the test in seconds. This score will be compared to the score obtained at baseline.
Assessment of cognitive status at 1 year using Trail Making Test | 1 year after surgery
  This test provides information visual search speed, scanning, speed of processing, mental flexibility, and executive functioning. The test is scored by the amount of time it takes to complete the test in seconds. This score will be compared to the scores obtained at baseline and 1 year after surgery.
Assessment of cognitive status at 3 months using the Digit Span | 3 months after surgery
  The Digit Span is used to measure the participant's memory span and number storage capacity. The scores range from 0-9 with 0 being short term memory impairment and 9 be no short term memory impairment. This score will be compared to the score obtained at baseline.
Assessment of cognitive status at 1 year using the Digit Span | 1 year after surgery
  The Digit Span is used to measure the participant's memory span and number storage capacity. The scores range from 0-9 with 0 being short term memory impairment and 9 be no short term memory impairment. This score will be compared to the scores obtained at baseline and 3 months after surgery.
Assessment of the cognitive status at 3 months using the Mini Mental Status Exam | 3 months after surgery
  The mini mental status exam measures cognitive impairment. Scores range from 0-30 with 0 being severe cognitive impairment and 30 being no cognitive impairment. This score will be compared to the score obtained at baseline.
Assessment of the cognitive status at 1 year using the Mini Mental Status Exam | 1 year after surgery
  The mini mental status exam measures cognitive impairment. Scores range from 0-30 with 0 being severe cognitive impairment and 30 being no cognitive impairment. The score obtained will be compared to the scores obtained at baseline and 3 months after surgery.
Assessment of cognitive status at 3 months after surgery using the Telephone Interview for Cognitive Status (TICS) | 3 months after surgery
  The telephone interview for cognitive status will only be used it the study team is unable to conduct the mini mental status exam in person. This test assesses cognitive function with scores ranging from 0-40 with 0 being severe cognitive impairment and 41 being no cognitive impairment.
Assessment of cognitive status at 1 year using the Telephone Interview for Cognitive Status (TICS) | 1 year after surgery
  The telephone interview for cognitive status will only be used it the study team is unable to conduct the mini mental status exam in person. This test assesses cognitive function with scores ranging from 0-40 with 0 being severe cognitive impairment and 41 being no cognitive impairment.
Maximum severity of delirium during hospital stay | Through the end of hospitalization, up to 3 months
  The patient will be assessed for delirium using the maximum total score on the Delirium Rating Scale-Revised 1998. The scale range is 0-32, with 0 being low delirium severity and 32 being high delirium severity.
Number of participants with hospital readmissions within 30 days of discharge | 30 days from hospital discharge
  Hospital readmissions will be measured.
Number of participants with emergency room visit within 30 days of hospital discharge | 30 days from hospital discharge
  Emergency Room Visits will be measured.
Number of days in hospital after surgery | Immediately after surgery until discharge, up to 3 months
  The number of days in hospital after surgery will be calculated for each patient.
Last pain score in the post-anesthesia care unit | Immediately before leaving the post-anesthesia care unit, up to 1 day
  The last pain score on the NRS pain scale of 0-10 taken in the post-anesthesia care unit by the post-anesthesia care unit staff. For this scale, 0 indicates no pain and 10 indicates the most severe pain.
Total morphine equivalents of opioids given in the post-anesthesia care unit | During post-anesthesia care unit stay, up to 1 week
  The total amount of opioids given to each patient in the post-anesthesia care unit will be converted to morphine equivalents for each patient.
Time first opioid given in the post-anesthesia care unit | The time the first opioid medication is given to the patient in the post-anesthesia care unit, up to 1 week
  The time will be noted when the first opioid is given to each participant in the post-anesthesia care unit.
Last pain score prior to hospital discharge | Immediately before hospital discharge
  The last pain score recorded for each participant on the NRS pain scale of 0-10. For this scale, 0 indicates no pain and 10 indicates the most severe pain.
Total amount of morphine equivalents during hospital stay | Duration of the hospital length of stay, up to 3 months
  The total amount of morphine equivalents will be measure for each participants hospital stay. The amount measured will be pro-rated tp the participant's length of stay.
The average pain score at 3 month follow-up | one week prior to end of 3 month follow-up
  The average pain score for each participant on the NRS pain scale of 0-10 over the week prior to the 3 month follow-up. These score are compared to scores from baseline assessments. For this scale, 0 indicates no pain and 10 indicates the most severe pain.
The average pain score at 12 month follow-up | one week prior to end of 12 month follow-up
  The average pain score for each participant on the NRS pain scale of 0-10 over the week prior to the 12 month follow-up. These score are compared to scores from baseline assessments. For this scale, 0 indicates no pain and 10 indicates the most severe pain.
Number of days with delirium | Duration of the hospital stay, up to 3 months
  The number of days with delirium will measured for each participant during the length of the hospital stay for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Charles C Edwards, MD, Principal Investigator — Mercy Hospital of Baltimore; Charles Brown, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown CH 4th, Jones EL, Lin C, Esmaili M, Gorashi Y, Skelton RA, Kaganov D, Colantuoni EA, Yanek LR, Neufeld KJ, Kamath V, Sieber FE, Dean CL, Edwards CC 2nd, Hogue CW. Shaping anesthetic techniques to reduce post-operative delirium (SHARP) study: a protocol for a prospective pragmatic randomized controlled trial to evaluate spinal anesthesia with targeted sedation compared with general anesthesia in older adults undergoing lumbar spine fusion surgery. BMC Anesthesiol. 2019 Oct 27;19(1):192. doi: 10.1186/s12871-019-0867-7. PMID 31656179